CLINICAL TRIAL: NCT06395181
Title: Effect of Whole Food Plant-based Diet in Patients with Obstructive Sleep Apnea
Brief Title: Whole Food Plant-based Diet Effect on Obstructive Sleep Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph Y. Cheung, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-011675
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea; Daytime Sleepiness
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diet Group: Whole Food Plant Based Diet (Experimental): Subjects with follow a whole food plant-based diet for 8 weeks.
  Interventions: Behavioral: Whole Food Plant-Based Diet
- Control Group: Usual Care (No Intervention): Subjects will not change their diet for 8 weeks.

INTERVENTIONS:
Behavioral: Whole Food Plant-Based Diet — A whole food, plant-based diet focuses on whole foods that are not processed. The diet places an emphasis on plant foods that are naturally lower in fat and includes eating a variety of plant foods (fruits, vegetables, beans and legumes, whole grains, nuts and seeds, spices and herbs).
  Other Names: WFPB Diet
  Arms: Diet Group: Whole Food Plant Based Diet

SUMMARY:
This research aims to develop a better understanding and clinical knowledge of the effects of a plant based diet on severity and daytime sleepiness in Obstructive Sleep Apnea.

ELIGIBILITY:
Inclusion Criteria:

* Daytime sleepiness with ESS score ≥ 5.
* Patient's prior sleep study with AHI between ≥ 10 and ≤ 45 (4% scoring criterion).
* On treatment for OSA, failed or not willing to use all other OSA treatment options
* Has access to a weight scale at home or able to come into the Sleep Clinic to be weighed after the 8-week plant-based diet period.

Exclusion Criteria:

* Pregnancy or lactation.
* Current use of a vegan diet.
* BMI ≤ 22.
* Complex, central sleep apnea.
* Pre-existing significant degree of cardio-pulmonary disease-heart failure with reduced EF of 35 or lower, unstable arrythmia, severe degree of pulmonary hypertension, severe degree of obstructive or restrictive lung disease including COPD and Interstitial lung disease.
* On weight loss medications or starting new exercise regimen during the 8-week plant-based diet period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in daytime sleepiness | Baseline, 8 weeks
  Measured using The Epworth sleepiness scale (ESS) which is an 8-item questionnaire that measures daytime sleepiness in participants. Possible scores range from 0-24, with higher scores indicating a higher average sleep propensity in daily life, and a worse outcome.
Change in Apnea-Hypopnea Index (AHI) | Baseline, 8 weeks
  Measured using the WatchPat One for at Home Sleep Apnea Test (HSAT), the Apnea-Hypopnea Index (AHI) assess severity of sleep apnea by counting apnea events during sleep. Normal range is less than 5 events per hour and severe is considered more than 30 events per hour.

SECONDARY OUTCOMES:
Change in weight | Baseline, 8 weeks
  Measured in kilograms (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheung, MD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials